CLINICAL TRIAL: NCT01887990
Title: Treatment of Suicidal Ideation With Intravenous Ketamine Infusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Dr. Richard Shelton, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: F120307001
Record Dates: First submitted 2012-08-07; First posted 2013-06-27 (Estimated); Results first posted 2015-07-09 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-04

CONDITIONS: Depression; Suicidal Ideation
MeSH Terms: conditions — Depression; Suicidal Ideation | interventions — Ketamine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Suicidal, Depression with Ketamine (Active Comparator): suicidal ideation and depression (no substance use disorder) 0.2 mg/kg IV ketamine administered as a one time dose
  Interventions: Drug: Ketamine
- Suicidal, Depression with Saline (Placebo Comparator): Suicidal ideation and depression (no substance use disorder) comparable amount of placebo (saline)
  Interventions: Drug: placebo
- Suicidal, opioid use with ketamine (Active Comparator): suicidal ideation,depression, opioid use disorder 0.2 mg/kg IV ketamine one time dose
  Interventions: Drug: Ketamine
- Suicidal, opioid use with Saline (Placebo Comparator): Patients with suicidal ideation and depression with opioid use disorder who are given comparable amount of placebo (saline) as would have been used with the Ketamine arm
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Ketamine — single dose IV 0.2 mg/kg ketamine
  Arms: Suicidal, Depression with Ketamine; Suicidal, opioid use with ketamine
Drug: placebo — saline infusion
  Other Names: saline
  Arms: Suicidal, Depression with Saline; Suicidal, opioid use with Saline

SUMMARY:
This study is dedicated to achieving better treatments for suicidal thoughts. Specifically, the investigators are studying the effect of a medication called ketamine to quickly treat suicidal thoughts and depression.

DETAILED DESCRIPTION:
This study is dedicated to achieving better treatments for suicidal thoughts. Specifically, we are studying the effect of a medication called ketamine to quickly treat suicidal thoughts and depression. Patients will be asked to participate in a research study to study how the use of a medication, ketamine, decreases your suicidal thoughts and improves their symptoms of depression. Ketamine is approved by FDA for use at higher doses in anesthesia, and recent clinical research suggests that it might benefit patients with major depressive disorder and suicidal thoughts. During clinical trials with over 10,000 patients, ketamine was proved to be safe as an anesthetic and studies with hundreds of patients with depression have demonstrated safety and lack of lasting side effects. This is a pilot study to test a new use of ketamine: treatment of suicidal thoughts. The study medication will be given in addition to usual psychiatric care.

ELIGIBILITY:
Inclusion Criteria:

1. Age : 19-64
2. Significant suicidality score on the Columbia Suicide Severity Rating Scale (C-SSRS)
3. Willing and able to provide informed consent.
4. Individuals with current substance abuse are allowed

Exclusion Criteria:

1. Pregnant or lactating; women of reproductive potential must have a negative urine pregnancy test (urine dipstick method)
2. Post-Partum state : defined as being within 2 months of delivery or miscarriage
3. Homicide risk as determined by clinical interview
4. Treatment with any medication known to specifically target the glutamate-NMDA receptor system (ie lamotrigine, acamprosate, memantine, riluzole or lithium)
5. Any known hypersensitivity or serious adverse effect associated with ketamine treatment.
6. Any clinically significant medical condition or therapy that would preclude treatment with ketamine, to include recent myocardial infarction or unstable angina
7. Medically unstable, including acute withdrawal from alcohol or benzodiazepines requiring the use of benzodiazepine treatment.
8. Any of the following DSM-IV diagnoses or categories:

   * Any current psychosis or history of a non-mood psychotic disorder (e.g., schizophrenia)
   * Currently in a manic or mixed episode
   * Current use (defined by urine dipstick test) or abuse of hallucinogenic drugs (except marijuana) such as phencyclidine
   * Any dissociative disorder
   * Any pervasive developmental disorder (e.g., autism)
   * A cognitive disorder (e.g., Alzheimer's Disease)
   * Cluster A personality disorder (e.g., schizoid or schizotypal); note that cluster B and C personality disorders may be included
   * Any eating disorder

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl B McCullumsmith, MD PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama Birmingham, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Suicidal, Depression With Ketamine: 0.2 mg/kg IV ketamine administered as a one time dose in patients with suicidal ideatin and depression without substance use
  Ketamine
- Suicidal, Depression With Saline: comparable amount of placebo (saline) as would have been used with the Ketamine arm
  placebo
- Suicidal, Depression and Opioid Use With Ketamine: suicidal, depressed with opioid use, given 0.2 mg/kg ketamine one time dose IV infusion
- Suicidal, Depression With Opioid Use With Saline: suicidal, depression with opioid use, given saline IV
Period: Overall Study
Arm/Group | Suicidal, Depression With Ketamine | Suicidal, Depression With Saline | Suicidal, Depression and Opioid Use With Ketamine | Suicidal, Depression With Opioid Use With Saline
Started | 7 | 7 | 2 | 2
Completed | 7 | 7 | 2 | 2
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Suicidal, Depression With Ketamine: suicidal and depressed, no substance use 0.2 mg/kg IV ketamine administered as a one time dose
  Ketamine
- Suicidal, Depression With Saline: suicidal and depressed, no substance use comparable amount of placebo (saline) as would have been used with the Ketamine arm
  placebo
- Suicidal, Depression and Opioid Use With Ketamine: suicidal and depressed, opioid use 0.2 mg/kg IV ketamine administered as a one time dose
  Ketamine
- Suicidal, Depression and Opioid Use With Ketamine: suicidal and depressed,opioid use comparable amount of placebo (saline) as would have been used with the Ketamine arm
  placebo
- Total: Total of all reporting groups
Arm/Group | Suicidal, Depression With Ketamine | Suicidal, Depression With Saline | Suicidal, Depression and Opioid Use With Ketamine | Suicidal, Depression and Opioid Use With Ketamine | Total
Number analyzed (Participants) | 7 | 7 | 2 | 2 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 37 (10) | 37 (11) | 31 (1) | 31 (4) | 35 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 0 | 0 | 6
  Male | 4 | 4 | 2 | 2 | 12
Region of Enrollment [Number; unit: participants]
  United States | 7 | 7 | 2 | 2 | 18

OUTCOME MEASURES:

1. Primary Outcome: Suicidality
Description: Scales and questionnaires using the Beck Scale for Suicidal Ideation. The Beck Scale is a self-report questionnaire. The items on this scale identify the presence and severity of suicidal ideation.
  Beck Scale for Suicidal Ideation has 19 items,preceded by a 5 item screener. Each item is rated on a 3 point scale from 0 to 2. Scores range from 0 to 48. Total scoreScores of 0 - 16 indicate low risk for suicide; scores of 16 or greater indicate higher risk for suicide.
Time Frame: 2 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Suicidal, Depression With Ketamine: 0.2 mg/kg IV ketamine administered as a one time dose
  Ketamine
Arm/Group | Suicidal, Depression With Ketamine | Suicidal, Depression With Saline | Suicidal, Opioid Use With Ketamine | Suicidal, Opioid Use With Saline
Number analyzed (Participants) | 7 | 7 | 2 | 2
units on a scale | 7.3 (11.4) | 21.5 (14.7) | 18.0 (25.5) | 0 (0)

2. Secondary Outcome: Depression
Description: Scales and Questionnaire using the MADRS (Montgomery-Asberg Depression Rating Scale) . This is a ten item diagnostic questionnaire used to measure the severity of depressive episodes in patients with mood disorders. the scale: 0 - 6 (normal/symptom absent), 7 - 19 (mild depression), 20 - 34 (moderate depression), and > 34 (severe depression).The overall score ranges from 0 to 60
Time Frame: 2 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Suicidal, Opioid Use With Ketamine: suicidal pts who have used opioids, in the ketamine treatment arm
- Suicidal, Opioid Use With Saline: suicidal patients who use opioids who received saline infusion or placebo
Arm/Group | Suicidal, Depression With Ketamine | Suicidal, Depression With Saline | Suicidal, Opioid Use With Ketamine | Suicidal, Opioid Use With Saline
Number analyzed (Participants) | 7 | 7 | 2 | 2
units on a scale | 43.9 (26) | 59.4 (17.2) | 22.5 (17.7) | 12.5 (3.5)

ADVERSE EVENTS:
Time Frame: 2 weeks
Groups:
- Suicidal, Depression With Ketamine: Suicidal with depression and no substance use 0.2 mg/kg IV ketamine administered as a one time dose
  Ketamine
- Suicidal, Depression With Saline: Suicidal with depression and no substance use comparable amount of placebo (saline) as would have been used with the Ketamine arm
  placebo
- Suicidal, Depression and Opioid Use With Ketamine: Suicidal with depression and opioid use 0.2 mg/kg IV ketamine administered as a one time dose
  Ketamine
- Suicidal, Depression and Opioid With Saline: Suicidal with depression and opioid use comparable amount of placebo (saline) as would have been used with the Ketamine arm
  placebo
Arm/Group | Suicidal, Depression With Ketamine | Suicidal, Depression With Saline | Suicidal, Depression and Opioid Use With Ketamine | Suicidal, Depression and Opioid With Saline
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 1/7 | 0/7 | 0/2 | 0/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Suicidal, Depression With Ketamine (N=7) | Suicidal, Depression With Saline (N=7) | Suicidal, Depression and Opioid Use With Ketamine (N=2) | Suicidal, Depression and Opioid With Saline (N=2)
sedation (Nervous system disorders) | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
short term followup small sample size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes